CLINICAL TRIAL: NCT05958485
Title: Glioblastoma Multiforme Patients in Clinical Trials: An Examination of Their Clinical Trial Experiences
Brief Title: A Close Examination of Patient Experiences in Glioblastoma Multiforme Clinical Research
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 82196870
Record Dates: First submitted 2023-07-14; First posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Glioblastoma Multiforme
Keywords: glioblastoma multiforme
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Clinical research can sometimes favor certain demographic groups. Additionally, there is limited research that delves into the factors that influence participation in clinical study, both positive and negative.

The goal is to identify the obstacles and challenges that prevent participation in glioblastoma multiforme clinical study, as well as the reasons for withdrawal or discontinuation.

Insights gained from this study will ultimately benefit those with glioblastoma multiforme who may be invited to participate in clinical trial in the years to come.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of glioblastoma multiforme
* No prior treatment for glioblastoma multiforme
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Female patients who are currently pregnant or nursing
* Enrolled in another research study
* Patients who are currently receiving any other investigational drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with glioblastoma multiforme who are actively considering participating in an observational clinical study, but have not yet completed enrollment and randomization.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Rate of patients who decide to enroll in a glioblastoma multiforme clinical study. | 3 months
Number of glioblastoma multiforme study participants who remain in clinical trial until completion. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Michaelsen SR, Christensen IJ, Grunnet K, Stockhausen MT, Broholm H, Kosteljanetz M, Poulsen HS. Clinical variables serve as prognostic factors in a model for survival from glioblastoma multiforme: an observational study of a cohort of consecutive non-selected patients from a single institution. BMC Cancer. 2013 Sep 3;13:402. doi: 10.1186/1471-2407-13-402. PMID 24004722
- [Background] Tosoni A, Gatto L, Franceschi E, Di Nunno V, Lodi R, Mura A, Di Battista M, Bartolini S, Brandes AA. Association between socioeconomic status and survival in glioblastoma: An Italian single-centre prospective observational study. Eur J Cancer. 2021 Mar;145:171-178. doi: 10.1016/j.ejca.2020.12.027. Epub 2021 Jan 22. PMID 33486440
- [Background] Ruda R, Bruno F, Pellerino A, Pronello E, Palmiero R, Bertero L, Crasto S, Polo V, Vitaliani R, Trincia E, Interno V, Porta C, Soffietti R. Observational real-life study on regorafenib in recurrent glioblastoma: does dose reduction reduce toxicity while maintaining the efficacy? J Neurooncol. 2022 Nov;160(2):389-402. doi: 10.1007/s11060-022-04155-9. Epub 2022 Oct 30. PMID 36309895

DOCUMENTS (1):
  • Informed Consent Form (2023-07-14): https://cdn.clinicaltrials.gov/large-docs/85/NCT05958485/ICF_000.pdf